CLINICAL TRIAL: NCT00352976
Title: Total Body Irradiation Dose De-escalation Study in Patients With Fanconi Anemia Undergoing Alternate Donor Hematopoietic Cell Transplantation
Brief Title: TBI Dose De-escalation for Fanconi Anemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2006-05; 0605M85788 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Fanconi Anemia
Keywords: Bone Marrow transplant; stem cell transplant; cord blood transplant; total body irradiation; thymic shielding
MeSH Terms: conditions — Fanconi Anemia | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Radiotherapy; Bone Marrow Transplantation; Stem Cell Transplantation; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with TBI (Experimental): Patients treated with total body irradiation, Fludarabine, Cyclophosphamide, Bone Marrow Transplantation, Mycophenolate Mofetil, and Sirolimus.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Total Body Irradiation; Procedure: Bone Marrow Transplantation; Drug: Mycophenolate Mofetil; Drug: Sirolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Day -5 through Day -2, subjects will receive chemotherapy of Cyclophosphamide via central line (i.e. Hickman or Broviac),10 mg/kg intravenously (IV)
  Other Names: cytoxan
Drug: Fludarabine — Day -5 through Day -2 prior to transplant; subjects will receive chemotherapy of Fludarabine via central line (i.e. Hickman or Broviac),35 mg/m^2 intravenous (IV)
  Other Names: fludara
Procedure: Total Body Irradiation — total body irradiation (300 cGy) with thymic shielding will be given six days before the stem cells are given (day -6). Thymic shielding is done by placing a piece of lead on the chest during the irradiation treatment so that the irradiation beams do not go to the thymus.
  Other Names: Radiation Therapy, Therapeutic radiation
Procedure: Bone Marrow Transplantation — A target of 5 * 10^6/kg and a minimum of 4 * 10^6 CD34+ cell/kg recipient weight will be collected by apheresis and used for transplant. In most cases this dose will be recovered in a single apheresis; however, a second or rarely third apheresis performed on the following days may be required to achieve the minimum dose.
  Other Names: Stem Cell transplantation
Drug: Mycophenolate Mofetil — Patients will receive MMF therapy beginning on day -3 through day +30 or for 7 days after engraftment, whichever day is later, if no acute graft-versus-host disease (GVHD). Engraftment is defined as 1st day of 3 consecutive days of absolute neutrophil count [ANC] > 0.5 * 10^9/L. MMF will be given at a dose of 15 mg/kg/dose every 8 hours by mouth(to a maximum dose of 1 gram).
  Other Names: MMF
Drug: Sirolimus — Sirolimus will be administered starting at day -3 with 8mg-12mg mg oral loading dose followed by single dose 4 mg/day with a target serum concentration of 3 to 12 mg/mL by high-performance liquid chromatography (HPLC). Levels are to be monitored 3 times/week in the first 2 weeks, weekly until day +60, and as clinically indicated until day +100 post-transplantation. In the absence of acute GVHD sirolimus may be tapered starting at day +100 and eliminated by day +180 post-transplantation.
  Other Names: Rapamycin

SUMMARY:
This is a single arm, total body irradiation (TBI) trial. All patients will be prescribed TBI 300 cGy with the goal of evaluating secondary endpoints.

DETAILED DESCRIPTION:
Study Treatment: Patients will receive voriconazole (antifungal therapy) by mouth beginning 1 month prior to conditioning therapy, if possible. 1) The subject is to receive total body irradiation (300 cGy) with thymic shielding; it will be given six days before the stem cells are given (day -6). 2) Day -5 through Day -2, subjects will receive a chemotherapy regimen of Fludarabine and Cyclophosphamide via central line (i.e. Hickman or Broviac). Starting Day -3, patients will receive sirolimus therapy with a taper commencing on day +180 and also mycophenolate mofetil (MMF) through day +30 or for 7 days after engraftment, whichever day is later, if no acute graft-versus-host disease (GVHD). 4) If the subject is receiving bone marrow or "peripheral" stem cells (cells collected from the donor's arm via a cell separator), on the day of transplantation, the stem cells taken from the donor will be put into a machine which will separate the lymphocytes (the cells that cause graft-versus-host disease [GVHD]) from the stem cells. If the subject is receiving an umbilical cord blood, the lymphocytes will not be removed because the risk of GVHD is not as high. Otherwise all patients will receive the same treatment. The stem cells are given as an infusion into the subject's existing catheter over 1-2 hours on day 0.5. On the day after transplant (day +1) subjects will be given G-CSF to stimulate the growth of the transplanted cells. 6. While receiving treatment and until the subject's blood counts recover he/she will have daily blood tests, and several bone marrow biopsies and aspirates. After recovery, subjects will be seen once a month for a health assessment and blood tests until at least 3 months after the cells have been infused. Additional blood tests or assessments may be done as medically indicated.

ELIGIBILITY:
Inclusion Criteria:

Meeting the definition of standard risk or high risk Fanconi anemia as defined in the next two sections:

* Standard risk patients must be <18 years of age with a diagnosis of Fanconi anemia with aplastic anemia (AA), myelodysplastic syndrome without excess blasts, or high risk genotype as defined below:

  * Aplastic anemia is defined as having at least one of the following when not receiving growth factors or transfusions:

    * platelet count <20 * 10^9/L
    * ANC <5 * 10^8/L
    * Hemoglobin <8 g/dL
  * Myelodysplastic syndrome (MDS) with multilineage dysplasia with or without chromosomal anomalies
  * High risk genotype (e.g. IVS-4 or exon 14 FANCC mutations, or BRCA1 or 2 mutations)
* High risk patients must have one or more of the following high risk features:

  * Advanced MDS (≥ 5% blast) or acute leukemia
  * Require additional HSCT for graft failure
  * History at any time of systemic fungal or gram negative infection
  * Severe renal disease with a creatinine clearance <40 mL/min
  * Age > 18 years
* Very high risk patients must have Advanced MDS (≥ 5% blast) or acute leukemia after initial hematopoietic stem cell transplant (HSCT)
* Patients must have an appropriate source of stem cells. Patients and donors will be typed for HLA-A, B, C and DRB1 using high resolution molecular typing.
* Adequate major organ function including:

  * Cardiac: ejection fraction >45%
  * Hepatic: bilirubin, AST or ALT, ALP <5 x normal
  * Karnofsky performance status >70% or Lansky >50 (if < 16 years of age)
* Women of child-bearing age must be using adequate birth control and have a negative pregnancy test.
* Written consent.

Exclusion Criteria:

* Available HLA-genotypically identical related donor in standard risk patients.
* Active central nervous system (CNS) leukemia at time of study enrollment.
* History of squamous cell carcinoma of the head/neck/cervix within previous 2 years.
* Prior radiation therapy that prevents further total body irradiation (TBI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2006-05-18 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L MacMillan, M.D., Principal Investigator — University of Minnesota Medical Center
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] MacMillan ML, DeFor TE, Young JA, Dusenbery KE, Blazar BR, Slungaard A, Zierhut H, Weisdorf DJ, Wagner JE. Alternative donor hematopoietic cell transplantation for Fanconi anemia. Blood. 2015 Jun 11;125(24):3798-804. doi: 10.1182/blood-2015-02-626002. Epub 2015 Mar 30. PMID 25824692
- See also: Trial 4 listed in the article corresponds to this clinical trial. — https://www.ncbi.nlm.nih.gov/pubmed/25824692

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With TBI: Patients treated with total body irradiation 300 cGy, Fludarabine 35 mg/m^2 (over 30 minutes daily for 4 days for a total dose of 140 mg/m^2), Cyclophosphamide 10 mg/kg (2 hour infusion for 4 days for a total dose of 40 mg/kg), Bone Marrow Transplantation, Mycophenolate Mofetil 1 mg/kg(over 30 minutes every 12 hours for 5 days) , and Sirolimus.
Period: Overall Study
Arm/Group | Treatment With TBI
Started | 83
Completed | 83
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 66
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 80
  Argentina | 1
  Canada | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Neutrophil Recovery
Description: Number of participant with neutrophil recovery. Neutrophil recovery is defined as absolute neutrophil count ≥500/µL for three consecutive days
Time Frame: by day 42
Population: 1 patient not evaluable since deceased at day 5 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 82
Participants | 78

2. Secondary Outcome: Number of Participants Experiencing Grade ≥3 Regimen Related Toxicity
Description: Regimen related toxicities (RRT) include: significant hemorrhagic cystitis, pulmonary hemorrhage, interstitial pneumonitis, GI hemorrhage, renal failure, erythroderma, and severe hepatic veno-occlusive disease
Time Frame: by day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 71

3. Secondary Outcome: Number of Participants With Secondary Graft Failure at 100 Days
Description: Secondary Graft Rejection by day 100
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 4

4. Secondary Outcome: Number of Participants Experiencing Acute Graft-versus-host Disease (GVHD)
Description: Number of participants experiencing acute GVHD (all grades) by day 100
Time Frame: at 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 15

5. Secondary Outcome: Number of Participants Experiencing Chronic GVHD
Description: Number of participants experiencing chronic Graft Vs Host Disease by 1 year
Time Frame: at one year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 6

6. Secondary Outcome: Number of Participants Experiencing Overall Survival
Description: Number of participants experiencing overall survival by 1 year
Time Frame: at one year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 70

7. Secondary Outcome: Number of Participants Experiencing Infections by Day 100
Time Frame: by day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 53

8. Secondary Outcome: Number of Participants Experiencing Infections by Day 180
Time Frame: by day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 55

9. Secondary Outcome: Number of Participants Experiencing Infections by Day 365
Time Frame: by day 365
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
Participants | 56

10. Secondary Outcome: Average Immunoglobulin G (IgG) Levels as a Measure of Immune Reconstitution After Transplant, by 100 Days
Time Frame: by 100 days
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Treatment With TBI: Average IgG levels as a measure of immune reconstitution after transplant
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 550.6 (285.4)

11. Secondary Outcome: Average IgG Levels as a Measure of Immune Reconstitution After Transplant, by 180 Days
Time Frame: by 180 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 652.9 (305.8)

12. Secondary Outcome: Average IgG Levels as a Measure of Immune Reconstitution After Transplant by 365 Days
Time Frame: by 365 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 724.0 (258.0)

13. Secondary Outcome: Average IgA Levels as a Measure of Immune Reconstitution After Transplant by 100 Days
Time Frame: by 100 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 88.0 (59.9)

14. Secondary Outcome: Average IgA Levels as a Measure of Immune Reconstitution After Transplant by 180 Days
Time Frame: by 180 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 98.7 (48.8)

15. Secondary Outcome: Average IgA Levels as a Measure of Immune Reconstitution After Transplant by 365 Days
Time Frame: by 365 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 107.2 (57.0)

16. Secondary Outcome: Average IgM Levels as a Measure of Immune Reconstitution After Transplant by 100 Days
Time Frame: by 100 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 71.1 (84.2)

17. Secondary Outcome: Average IgM Levels as a Measure of Immune Reconstitution After Transplant by 180 Days
Time Frame: by 180 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 77.0 (60.3)

18. Secondary Outcome: Average IgM Levels as a Measure of Immune Reconstitution After Transplant by 365 Days
Time Frame: by 365 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With TBI
Number analyzed (Participants) | 83
mg/dL | 82.8 (57.9)

ADVERSE EVENTS:
Time Frame: Through after transplant by 365 Days
Arm/Group | Treatment With TBI
All-Cause Mortality (participants affected / at risk) | 13/83
Serious Adverse Events (participants affected / at risk) | 4/83
Other Adverse Events (participants affected / at risk) | 75/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With TBI (N=83)
Progressive Disease (Blood and lymphatic system disorders) | 1 (3)
Relapsed (Blood and lymphatic system disorders) | 1 (2)
Infection (Infections and infestations) | 2 (2)
Blood/Bone Marrow GVHD (Blood and lymphatic system disorders) | 1 (1)
Graft failure (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With TBI (N=83)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Injury, poisoning and procedural complications, other (Blood and lymphatic system disorders) | 1 (1)
Investigations, other (Blood and lymphatic system disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 3 (5)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
hemolysis (Blood and lymphatic system disorders) | 1 (1)
hypoatremia (Blood and lymphatic system disorders) | 1 (1)
neurotoxicity (Blood and lymphatic system disorders) | 1 (1)
cardiomegaly (Cardiac disorders) | 1 (1)
myringotomy (Ear and labyrinth disorders) | 1 (1)
Hemorrhage (Gastrointestinal disorders) | 1 (3)
Ileum obstruction (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
cholecystectomy (Gastrointestinal disorders) | 1 (1)
hepatic steatosis (Gastrointestinal disorders) | 1 (1)
hernia (Gastrointestinal disorders) | 1 (1)
ischemic hepatitis (Gastrointestinal disorders) | 1 (1)
pancreatic inflammation (Gastrointestinal disorders) | 1 (1)
proximal obstruction (Gastrointestinal disorders) | 1 (1)
multi-system failure (General disorders) | 3 (3)
Hemmorhage (Hepatobiliary disorders) | 1 (1)
Veno-Occlusive Disease (Hepatobiliary disorders) | 3 (4)
allergic reaction (Immune system disorders) | 1 (1)
Herpes (Infections and infestations) | 5 (6)
Infection (Infections and infestations) | 42 (122)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Engraftment Syndrome (Injury, poisoning and procedural complications) | 9 (9)
GI bleed (Injury, poisoning and procedural complications) | 13 (15)
Injury, poisoning and procedural complications, other (Injury, poisoning and procedural complications) | 2 (2)
Investigations, other (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Type 2 Diabetes (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 6 (6)
altered mental status (Nervous system disorders) | 1 (1)
intracranial hemorrhage (Nervous system disorders) | 2 (2)
neurotoxicity (Nervous system disorders) | 2 (3)
vision impairment (Nervous system disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 26 (30)
Dialysis (Renal and urinary disorders) | 6 (7)
Injury, poisoning and procedural complications, other (Renal and urinary disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug Toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intubation (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 31 (74)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respirtory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 7 (9)
bilateral interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
pnuemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary cytolytic thrombi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug Toxicity (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 24 (26)
Neuropathy (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
Hemorrhage (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 11 (13)
atrial fibrilation (Cardiac disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
cardiomyopathy (Cardiac disorders) | 1 (1)
edema (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT00352976/Prot_SAP_000.pdf